CLINICAL TRIAL: NCT06102148
Title: The Effect Of Proprioceptive Neuromuscular Facilitation Techniqueson Pain, Motor Functions, Fatique and Health Related Quality of Life in Patients With Multiple Sclerosis: A Randomized, Single-blind Study.
Brief Title: The Effect Of Proprioceptive Neuromuscular Facilitation Techniqueson in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilay Comuk Balci (Other)
Responsible Party: Sponsor-Investigator, Nilay Comuk Balci, Associate professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/413
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Proprioceptive Neuromuscular Facilitation; Pain; Motor Function; Fatigue; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Pain; Fatigue | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Group (Experimental)
  Interventions: Other: PNF Group
- Control Group (Sham Comparator)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: PNF Group — Exercise training and PNF training
  Arms: PNF Group
Other: Control Group — Exercise training
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effects of PNF techniques on pain, motor function, fatigue and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of Relapsing-Remitting MS (RRMS) as defined by McDonald criteria
* 18-65 years of age
* an Expanded Disability Status Scale (EDSS) score < 4
* relapse-free for the last 3 months
* cognitive impairment that was defined with mini mental test.

Exclusion Criteria:

* a history of different neurological diseases
* having any contraindication for exercise
* having orthopedic, vision, hearing, or perception problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | through study completion, an average of 1 year
  Pain
Multiple Sclerosis Quality of Life-54 (MSQoL-54) | through study completion, an average of 1 year
  Quality of Life
Fatigue Severity Scale and Fatigue Impact Scale (FIS) | through study completion, an average of 1 year
  Fatigue
Timed Up and Go (TUG) | through study completion, an average of 1 year
  Mobility and Balance
The Six-Minute Walk Test (6-MWT) | through study completion, an average of 1 year
  Functionality
Hand Dexterity | through study completion, an average of 1 year
  Hand Dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)